CLINICAL TRIAL: NCT05700942
Title: Transcutaneous Spinal Direct Current Stimulation to Enhance Locomotor Rehabilitation After Spinal Cord Injury
Brief Title: AMPLIFY Study: Transcutaneous Spinal Direct Current Stimulation to Enhance Locomotor Rehabilitation After SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Brooks Rehabilitation (Other); The Craig H. Neilsen Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202201350
Record Dates: First submitted 2022-09-19; First posted 2023-01-26 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Stratified randomization will be used to allocate participants to their treatment group (higher or lower dose of tsDCS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- High Dose Intervention (Experimental): tsDCS will be delivered to the lumbar region of the spinal cord during LT using a commercially available stimulation unit (Soterix Medical, Inc., New York, NY). tsDCS electrodes are comprised of a 10x5 cm carbon rubber electrode encased in a saline-soaked sponge. The anode electrode will be placed on the skin over the spinal processes of the 11th and 12th thoracic vertebrae, and the two cathode electrodes will be placed on each side of the umbilicus. For the high dose group, a standard dosage of 30 continuous minutes of 2.5 mA stimulus will be used.
  Interventions: Device: High Dose Intervention-tsDCS
- Low Dose Intervention (Active Comparator): tsDCS will be delivered to the lumbar region of the spinal cord during LT using a commercially available stimulation unit (Soterix Medical, Inc., New York, NY). tsDCS electrodes are comprised of a 10x5 cm carbon rubber electrode encased in a saline-soaked sponge. The anode electrode will be placed on the skin over the spinal processes of the 11th and 12th thoracic vertebrae, and the two cathode electrodes will be placed on each side of the umbilicus. The low dose condition will use an identical montage and stimulation arrangement, except the stimulation will be delivered briefly at the beginning and end of the stimulation period (30 seconds) with a three-second ramp.
  Interventions: Device: Low Dose Intervention-tsDCS

INTERVENTIONS:
Device: High Dose Intervention-tsDCS — Subjects will receive a high dose tsDCS (2.5mA, 30 mins) LT (4x/week, 5 weeks)
  Other Names: standardized locomotor training (LT)/ walking rehabilitation on treadmill and overground
  Arms: High Dose Intervention
Device: Low Dose Intervention-tsDCS — Subjects will receive a low dose tsDCS (2.5mA, 30 mins) LT (4xweek/ 5 weeks)
  Other Names: standardized locomotor training (LT)/ walking rehabilitation on treadmill and overground
  Arms: Low Dose Intervention

SUMMARY:
Locomotor training (LT) facilitates recovery of spinal locomotor networks after incomplete spinal cord injury (ISCI), but walking impairments persist. A limitation of LT is insufficient excitation of spinal locomotor circuits to induce neuroplastic recovery. Transcutaneous spinal direct current stimulation (tsDCS) is a non-invasive approach to increase spinal excitation and modulate spinal reflexes. The study will examine if tsDCS combined with LT enhances locomotor rehabilitation after ISCI.

DETAILED DESCRIPTION:
Transcutaneous spinal direct current stimulation (tsDCS) is a mild, non-invasive approach to increase spinal excitation and modulate spinal reflexes. Although ample evidence suggests tsDCS could enhance the effect of locomotor rehabilitation, the efficacy of this combinatorial strategy has not been investigated in individuals with ISCI. Based on supportive evidence from our prior feasibility study, the investigators will examine initial efficacy and mechanistic changes from combined tsDCS and locomotor training (tsDCS+LT).

Specific aim 1: To determine the effect size and variance of response to combined tsDCS and LT to enable power analysis for a larger clinical trial. Participants (chronic, motor ISCI) will complete a double-blind, randomized parallel-group design study to examine the effects of tsDCS (20 sessions, 30 minutes, anodal, 2.5 mA) delivered concurrently with LT. Walking outcomes will be measured pre- and post-intervention to compare the effects of tsDCS+LT versus sham+LT. Primary outcomes will be changes in overground walking speed and endurance.

Specific aim 2: To test the hypothesis that tsDCS+LT increases spinal motor excitability and reflex modulation. Spinal excitability will be assessed by Hoffman reflex amplitudes. Reflex modulation will be assessed by normalized measures of reflex post-activation depression as well as by gait phase-dependent modulation.

This proposed clinical trial will utilize a double-blind, randomized parallel-group experimental design. Once screening is complete, individuals will be enrolled for approximately two months to complete all study procedures. Participants will be randomized to receive either the higher or lower (sham) dose of tsDCS. The intervention will consist of 20 sessions (5 weeks x 4 sessions/week) of LT with the assigned tsDCS dose.

All participants will complete assessments at three time points. Clinical assessments to characterize injury severity and baseline characteristics, biomechanical, electromyographic (EMG) and clinical assessments of walking function, and reflex testing will be completed pre-intervention and one to three days post-intervention. A follow-up assessment consisting of clinical walking and mobility function outcomes only will be reassessed two weeks post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 65 years of age
* Single chronic SCI for ≥ 1 year classified as neurologic level T12 or above based on the International Standards for the Neurological Classification of SCI67 and classified according to the American Spinal Injury Association Impairment Scale (AIS) as motor incomplete (AIS C or D) at initial screening
* Medical stability with clearance from physician
* Ability to walk 3 meters with or without devices, braces, or assistance of one person
* Ability to provide informed consent.

Exclusion Criteria:

* Current diagnosis of an additional neurologic condition such as multiple sclerosis, Parkinson's disease, stroke, or brain injury
* Presence of unstable or uncontrolled medical conditions such as cardiovascular disease, myocardial infarction (<1 year prior), pulmonary infection or illness, renal disease, autonomic dysreflexia, infections, pain, heterotopic ossification
* Cognitive or communication impairments limiting communication with study staff or ability to provide informed consent
* Lower extremity joint contractures limiting the ability to stand upright and practice walking
* Skin lesions or wounds affecting participation in walking rehabilitation
* Acute or unstable fracture, diagnosis of osteoarthritis or bone impairments affecting safe participation in walking rehabilitation
* Severe spasticity or uncontrolled movements limiting participation in walking rehabilitation
* Body weight or height that is incompatible with safe use of a support harness and body weight support system
* Pain that limits walking or participation in walking rehabilitation
* Current participation in rehabilitation to address walking function
* Botox injections in lower extremity muscles affecting walking function within 4 months of study enrollment
* Legal blindness or severe visual impairment
* Known pregnancy
* Implanted metal hardware of the spine below the 8th thoracic vertebrae or in region of electrode placement
* Implanted cardiac pacemaker or baclofen pump

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in 10-Meter Walk Test (10MWT) | Baseline, Week 6, Week 8
  Is a performance measure used to assess walking speed in meters per second over a short distance. Performance assessment of comfortable and fastest safe walking speed for 10 meters. A reduced time (in seconds) to complete the 10-Meter Walk Test reflects improvement in walking function
Change in 6-Minute Walk Test (6MWT) | Baseline, Week 6, Week 8
  The distance that a patient should walk based on their height, weight, age, and gender. Performance assessment of walking endurance for 6 minutes. An increase in the number of meters walked during this assessment reflects an improvement in walking endurance.
Change in H-Reflex Post Activation Depression | Baseline, Week 6
  Assessment that quantifies the appropriate reduction in motor response to repeated sensory inputs. Increased post-activation depression (reduced motor response as measured with electromyography) reflects improved spinal modulation and may reflect normalization of an overactive stretch reflex.
Change in H-Reflex Gait Phase Modulation | Baseline, Week 6
  Assessment that quantifies the appropriate modulation of motor response to sensory input across the gait cycle. Improved modulation may reflect improved spinal rhythmic output to permit improved walking function.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Fox, DPT, PhD, Principal Investigator — University of Florida
Locations (1):
- Brooks Rehabilitation Hospital, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No